CLINICAL TRIAL: NCT06123819
Title: Correlation of Shear-wave Elastography Parameters With the Molecular Subtypes of Breast Cancer
Brief Title: Shear-wave Elastography in Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Walaa Gamal Abdelnasser, doctor, Assiut University
Other Study IDs: shear-wave in breast cancer
Record Dates: First submitted 2023-10-25; First posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Elasticity Imaging Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: elastography — . First, strain elastography (it is based upon the fact that hard tissue is more difficulty compressed than soft tissue. SE is a technique that measures the tissue deformation generated by compression, which may be applied with a probe on the body surface for static imaging) will be performed. The elastogram image of the detected lesion, will be evaluated Using color coding ranging from blue, through green and red. All lesions will be scored on elastogram in terms of their Stiffness compared to normal parenchyma. Second, shear wave elastography (is a method to generate shear waves and measure SWV ,based on the principle of fast propagation of shear wave speed in hard tissue and slow propagation in soft tissue , the hardness of tissue is indirectly reflected by measuring shear wave speed ) , will also be calculated individually.

SUMMARY:
The purpose of this study is to determine the relationship of the SWE elastic modulus and the molecular types of breast cancer .

DETAILED DESCRIPTION:
Breast cancer is the most common cancer of women world wide, and it is the second leading cause of death following lung cancer. Treatment options for breast cancer have changed in recent years; primary conventional surgery is no longer considered the most appropriate option for every patient.

The Age, molecular subtype, spread of the tumor, axillary lymph node status(as it is the first site to be metastasized by breast cancer through the lymphatic vessels) , and patient preference are the main determinants of breast cancer treatment, and a multidisciplinary approach is necessary.

With the development of molecular biology, it has been recognized that breast cancer has large biological diversity and high heterogeneity, which result in different morphological subtypes. According to immunehistochemical indexes such as estrogen receptor (ER), progesterone receptor (PR),proliferating cell nuclear antigen (Ki-67), and human epidermal growth factor receptor-2 (HER-2), clinicians determine 4 main molecular subtypes of breast cancer : -luminal A (ER+ or PR+, HER2-, andKi67 < 15%).

* luminal B (ER+ or PR+, HER2-/+,and Ki67 > 15%).
* triple negative (ER-, PR-, andHER2-).
* HER2+ (ER-, PR-, and HER2+). Determination of the molecular subtype of is the most important factor in systemic breast cancer treatment ; for example, it is generally preferred to use endocrine therapy in cases of hormone receptor positivity, anti-HER2 drugs in cases of human epidermal growth factor receptor2 (HER2) positivity, and chemotherapy in triple-negative patients.

The molecular subtype also determines recurrence and prognosis. For example, the triple negative subtype shows recurrence more frequently than other subtypes, while the luminal A subtype has a better prognosis.

Ultrasound (US) is an important modality for the detection and characterization of breast masses; it is also the first guiding method to be chosen for percutaneous biopsies in daily practice. Elastography is us based imaging modality recently developed to measure the elasticity of tissues using sound waves. Two-dimensional shear-wave elastography (SWE) is a newly emerging elastography technique, which can display tissue stiffness in a quantified form to obtain the biological information of the primary lesion . At present, many studies have verified the diagnostic value of SWE for benign and malignant lesions in breasts . The technique has been widely employed to check the thyroid, pancreas, kidney, prostate, liver, and other organs while few studies about axillary node metastasis (ANM) and its application for the molecular classification of breast cancer were reported .

The purpose of this study is to determine the relationship of the SWE elastic modulus and the molecular types of breast cancer .

ELIGIBILITY:
Inclusion Criteria:

* Women who were diagnosed with invasive breast cancer and did not receive neoadjuvant treatment and who previously did not have an operation on the same breast or axillary fossa .

Exclusion Criteria:

* Women who were diagnosed with non-invasive breast cancer and who receive neoadjuvant treatment and who previously had an operation on the same breast or axillary fossa .
* patients who expressed their oppositionto the use of their personal data.

Ages: 18 Years to 75 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Based on determining the main outcome variable ,the estimated minimum required sample size is 60 patients.
  The sample size was calculated using Epi-info version 7 software, based on the following assumptions:
  Main outcome variable is correlate various pattern of non mass lesions with histopathology for further management. Based on previos accuracy is 81%. Based on this percentage confidence limits of 6% and a confidence level=80%.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Changes in the tumor stiffness values on SWE were significantly associated with aggressive histopathologic features of breast cancer. | baseline
  We analyze 545 consecutive women (mean age, 52.7 ± 10.7 years; range, 26-83) with breast cancer who underwent preoperative breast ultrasound with SWE parameters (Emax, Emean, and Eratio) and the histopathologic information from surgical specimens including histologic type, histologic grade, size of invasive cancer, hormone receptor and HER2 status, Ki-67 proliferation index, and axillary LN status were analyzed. The relationships between SWE parameters and histopathologic findings were analyzed using an independent sample t-test, one-way ANOVA test with Tukey's post hoc test, andlogistic regression analyses.

CONTACTS AND LOCATIONS:
Overall Officials: sherin ezzat, Study Director — Assiut University

REFERENCES:
- [Background] Gweon HM, Youk JH, Son EJ, Kim JA. Clinical application of qualitative assessment for breast masses in shear-wave elastography. Eur J Radiol. 2013 Nov;82(11):e680-5. doi: 10.1016/j.ejrad.2013.08.004. Epub 2013 Aug 14. PMID 23988689
- [Background] Yoon JH, Ko KH, Jung HK, Lee JT. Qualitative pattern classification of shear wave elastography for breast masses: how it correlates to quantitative measurements. Eur J Radiol. 2013 Dec;82(12):2199-204. doi: 10.1016/j.ejrad.2013.08.047. Epub 2013 Sep 3. PMID 24041435